CLINICAL TRIAL: NCT06605716
Title: Assessing the Frequency of Trigeminocardiac Reflex in Maxillary and Mandibular Cyst Operations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Bedreddin Cavlı, Assistant Professor Doctor, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: KutahyaHSU/BedreddinCavli/002
Record Dates: First submitted 2024-07-08; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Trigeminocardiac Reflex; Jaw Cysts; Hemodynamic Instability
Keywords: Trigemino-Cardiac Reflex; Jaw cysts; Hemodynamic instability,
MeSH Terms: conditions — Jaw Cysts

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maxilla (Experimental): Presence of cystic structures larger than 1 cm in the maxilla with a surgical indication for enucleation Healthy adults
  Interventions: Procedure: Enucleation of cysts
- Mandibula (Experimental): Presence of cystic structures larger than 1 cm in the mandible with a surgical indication for enucleation Healthy adults
  Interventions: Procedure: Enucleation of cysts

INTERVENTIONS:
Procedure: Enucleation of cysts — Surgical removal of cystic structures larger than 1 cm in patients included in the study arms. Patients were monitored for TCR during the procedure.

SUMMARY:
The goal of this clinical trial is to investigate the frequency of trigeminocardiac reflex development during the surgical removal of large cystic structures within the maxillary and mandibular bones in healthy adults. The main questions it aims to answer are:

* What is the frequency of trigeminocardiac reflex development during the related surgical procedure?
* Does the frequency of TCR differ between the maxilla and mandible?
* Does the risk level for TCR increase in surgical procedures near vital structures (sinus floor, nasal floor, inferior alveolar nerve) depending on the size of the cyst?

DETAILED DESCRIPTION:
A total of 34 patients, including 17 undergoing maxillary and 17 undergoing mandibular cyst enucleations, were included in the study. Evaluation of the patients was performed using orthopantomogram films. The distances of the relevant cysts from surrounding vital structures were recorded, confirmed, and documented as necessary with cone beam computed tomography images if less than or greater than 1 mm.

Patients were divided into 2 groups, evenly comprising 17 patients each in maxilla and mandible groups. The surgeries included in the study were performed by a single surgeon. Surgical procedures utilized crestal incisions with horizontal and vertical relaxing incisions related to the size of the cysts.

The follow-up of the trigeminocardiac reflex (TKR) was conducted due to the occurrence of sudden bradycardia that was unprecedented following a tachycardia, which could develop within a few seconds and showed improvement when the procedure was paused. To ensure accurate and timely monitoring of this sudden process and to track potential asystole, patients were preferred to be monitored. Monitoring was facilitated using 5-channel Contec Medical Systems (Hebei, China) monitors. Throughout the procedure, heart rate, systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure, and oxygen saturation were recorded.

The records were obtained during 6 separate surgical stages: firstly, during local anesthesia application; subsequently, during incision, flap elevation, removal of the bone barrier, manipulation and extraction of the cyst, irrigation, and suturing stages. Sudden changes occurring during the procedure were recorded along with their timing.

In defining TCR (Trigeminocardiac Reflex) in the literature, various reference measurement methods include sudden drops in heart rate by more than 10%, more than 20%, or dropping below 60 beats per minute. To highlight these different proportional reference drop values, severity grading was used in the observed TCR findings. Sudden drops in heart rate between 10% and 20% were classified as mild TCR (TKR-1), drops exceeding 20% and heart rate falling below 60 bpm as moderate TCR (TKR-2), and the presence of asystole, syncope, or need for atropine application as severe TCR (TCR-3). The total TCR across all grades was termed as t-TCR. TCR calculation was based on heart rate measurements taken at the beginning of each surgical stage.

To exclude vasovagal syncope, commonly cited as the most frequent cause of neurological emergencies, and high anxiety as etiological factors, patients initially underwent anxiety assessments. Individuals with high anxiety levels were excluded from the study. Patients' anxiety levels were assessed using the Amsterdam Preoperative Anxiety and Information Scale (APAIS) and the State-Trait Anxiety Inventory-State (STAI-S).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients with cystic lesions at least 1 cm in diameter in the maxilla and mandible
* Patients with no systemic health problems

Exclusion Criteria:

* Pregnant or breastfeeding female patients
* Patients with systemic health problems
* Patients with mental or neurological disorders
* Patients taking antidepressants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Heart rate monitoring | During the operation
  All patients in all research arms monitored prior to enucleation of cystic structures in the maxilla and mandible had their heart rate monitored throughout the procedure.
Systolic, and diastolic blood pressure monitoring | During the operation
  All patients in all research arms monitored prior to enucleation of cystic structures in the maxilla and mandible had their systolic, and diastolic blood pressure monitored throughout the procedure.
Oxygen saturation monitoring | During the operation
  All patients in all research arms monitored prior to enucleation of cystic structures in the maxilla and mandible had their oxygen saturation monitored throughout the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Bedreddin Cavlı, Asst Prof, Principal Investigator — Kutahya University of Health Sciences, Faculty of Dentistry
Locations (1):
- Kutahya University of Health Sciences, Kütahya, Turkey (Türkiye)

DOCUMENTS (1):
  • Study Protocol (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT06605716/Prot_000.pdf